CLINICAL TRIAL: NCT00999180
Title: Botulinum Toxin Type A and Kinesitherapy Use in the Functional Performance of Post-stroke Patients
Brief Title: Botulinum Toxin Type A and Kinesitherapy of Post-stroke Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Ailton de Souza Melo, Botulinum Toxin Type A and Kinesitherapy Use in the Functional Performance of Post-stroke Patients, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UFBA-064
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2009-10

CONDITIONS: Stroke
Keywords: Botulinum Toxin; Rehabilitation; Stroke
MeSH Terms: conditions — Stroke | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Btx-A and Kinesiotherapy (Active Comparator): The botulinum toxin group will have the syringe filled with botulinum toxin type A (Dysport). During this period the patients will be followed by the IBR facility where will undergo a protocol of physical therapy comprising muscle strengthen, flexibility, endurance, and functional training.
  Interventions: Procedure: Botulinum toxin type A and kinesiotherapy
- Saline and Kinesiotherapy (Placebo Comparator): The control group will have the syringe filled with saline.During this period the patients will be followed by the IBR facility where will undergo a protocol of physical therapy comprising muscle strengthen, flexibility, endurance, and functional training.
  Interventions: Procedure: Saline and Kinesiotherapy

INTERVENTIONS:
Procedure: Botulinum toxin type A and kinesiotherapy — Stroke, Botulinum Toxin
  Other Names: Dysport
  Arms: Btx-A and Kinesiotherapy
Procedure: Saline and Kinesiotherapy — Saline and Kinesiotherapy
  Arms: Saline and Kinesiotherapy

SUMMARY:
The objective of this study is to assess if the association of botulinum toxin type A and kinesitherapy is superior to kinesitherapy and 0,9% saline for the functional performance in post-stroke patients.

Hypothesis H(0): BT-A associated to kinesitherapy is not superior to kinesitherapy in the function of hemiparetic post-stroke patients.

H(1): BT-A associated to kinesitherapy is superior to kinesitherapy in the function of hemiparetic post-stroke patients.

DETAILED DESCRIPTION:
The patients will be oriented regarding to the study steps and potential risks of the procedures. They will be assessed by a spasticity-experienced physical therapist. Demographical data will be collected by a questionnaire, the range of movement will be measured with a goniometer, and the muscle tone will be determine by the modified Ashworth scale, with the patient in dorsal decubitus. The presence of hypertonia equal or superior to 2 will assign the respective muscle to injection. Then the patients will be conducted to another room, where another therapist will assess the functional performance by the "timed up and go" (TUG) test, a six-minutes duration walking, and the Fugl-Meyer scale for the upper limb, with the patient in the seated position. During the TUG test the patient is asked to stand up from a chair and walk 3 meters, turn around 180 degrees, and walk back to the chair, assuming 10 seconds as the normal. The 6 minutes walking test will measure the distance in meters in a previously demarcated place. A staff will constantly stimulate the patient verbally, to walk as fast as possible.

Posteriorly the patients will be set in another room, where a neurologist will inject one of the two possible substances, with a pre-determined dosage and dilution. The botulinum toxin group will have the syringe filled with botulinum toxin type A (Dysport) and the control group will have the syringe filled with saline. All the patients will be reassessed in three and six months for a new injection, and will undergo the last evaluation in nine months.

During this period the patients will be followed by the IBR facility where will undergo a protocol of physical therapy comprising muscle strengthen, flexibility, endurance, and functional training (appendix D). There will be appointments twice a week, one day apart. The duration of the session will be 30 minutes, being 1 minute the interval between the activities. The first 5 minutes will comprise the flexibility exercises, with sustained stretching (15 seconds) and joint mobilizations, followed by a muscle strength exercise involving concentric and eccentric movements, with a progressive charge depending on the patient performance within the following 10 minutes. The last 15 minutes will have a functional training involving gait and upper limb activity combined with endurance training. These activities will be divided into two days: the first day for the trunk and upper limb, and the second for the pelvic, gait, and lower limb exercises. This protocol will be carried out by two physical therapist blinded regarding to the drug injection.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cerebrovascular accident and indication for the botulinum toxin injection (Hypertonia equal or superior to 2 according to the Ashworth scale).
* Patients followed by the physical therapy staff at the IBR and HAS, with 2 appointments per week.
* Patients from both sexes with ages superior to 18 years
* To have the minimum of one a maximum of five years post post-stroke.

Exclusion Criteria:

* Patients with age superior to 70 years
* Cognitive impairment
* Poorly controlled arterial hypertension
* Presence of joint blockade
* Unable to walk independently
* Use of orthesis as a gait aid
* Use of botulinum toxin within the last six months
* Use of systemic drugs for reduction of tonus
* Blood, liver, or kidney disorders and pregnant or lactating women
* Cardiopathy
* Comprehension aphasia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-03 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Functional performance assessed by TUG test and six minutes walking: an improvement of more than 50% of the expected for each test. | one year

SECONDARY OUTCOMES:
Muscle tone: a reduction of at least 1 point in the Ashworth scale. Range of movement: an improvement of at least 10 degrees. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ailton Melo, PHD, Principal Investigator — Federal University of Bahia
Locations (1):
- Federal University of Bahia, Salvador, Estado de Bahia, Brazil